CLINICAL TRIAL: NCT00449761
Title: A Phase II, Multicentre Study of Oral LBH589 in Patients With Accelerated Phase or Blast Phase (Blast Crisis) Chronic Myeloid Leukemia With Resistant Disease Following Treatment With at Least Two BCR-ABL Tyrosine Kinase Inhibitors
Brief Title: Efficacy and Safety of LBH589B in Adult Patients With Refractory Chronic Myeloid Leukemia in Accelerated or Blast Phase
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2211
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: Refractory; Chronic Myeloid; Leukemia; accelerated phase; blast phase (blast crisis); adults; oral LBH589
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Blast Crisis | interventions — Panobinostat

ARMS (1):
- Panobinostat (Experimental): Participants received panobinostat 20 milligrams (mg) orally once daily (OD), three times a week as part of a 4 week (28 day) treatment cycle. Panobinostat was administered at the same time each morning, and with an 8oz/240 milliliter (ml) of water after a fasting period of at least two hours (water was allowed). Participants could continue this treatment until an unacceptable toxicity that precludes further treatment was experienced, or until disease progression.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat

SUMMARY:
This study will evaluate the efficacy and safety of LBH589B in adult patients with chronic myeloid leukemia who are in accelerated phase or blast phase (blast crisis) with resistant disease following treatment with at least two BCR-ABL tyrosine kinase inhibitors

DETAILED DESCRIPTION:
study was designed to assess the hematologic response associated with treatment of oral panobinostat. Hematologic response is defined as the overall of complete hematologic response (CHR), and of no evidence of leukemia (NEL) and of the return to chronic phase (RTC). Hematologic responses were to be confirmed after 4 weeks, and all criteria listed below for each type of response were to be concomitantly met to result into a response.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged ≥ 18 years old
* Diagnosis of Philadelphia chromosome positive accelerated or blast phase chronic myeloid leukemia defined as:

Accelerated phase - the presence of at least one of the following:

* ≥15% but <30% blasts in blood or bone marrow
* ≥30% blasts plus promyelocytes in peripheral blood or bone marrow (providing that <30% blasts present in bone marrow)
* ≥ 20% basophiles in the peripheral blood
* Thrombocytopenia <100 X 109 /L unrelated to sole therapy

Blast phase (blast crisis) - the presence of one of the following:

* ≥ 30% blasts in the blood, in bone marrow or both
* Extramedullary infiltrates of leukemic cells other than liver or spleen involvement
* Prior treatment with at least two a fusion gene of the BCR and ABL genes (BCR-ABL) tyrosine kinase inhibitors (i.e., imatinib, nilotinib, or dasatinib) and demonstrated resistance to the most recent kinase inhibitor therapy. Resistance to a BCR-ABL tyrosine kinase inhibitors (TKI) for this study was defined as:

  * Progression from chronic phase to either accelerated phase or blast crisis
  * Progression from accelerated phase to blast crisis
  * No hematologic response (defined as not achieving complete hematologic response (CHR), no evidence of leukemia (NEL) or return to chronic phase (RTC)) within 3 months of starting therapy
  * Increasing blast counts in peripheral blood of increasing marrow leukemic infiltrate (MLI, the percent marrow blasts multiplied by marrow cellularity)
* Patients with a history of intolerance to one BCR-ABL kinase inhibitors (defined as discontinuation of treatment due grade 3 or 4 adverse events related to treatment) will be considered eligible to enter the study if they demonstrate resistance to their most recent BCR-ABL kinase inhibitor. Intolerance was defined as discontinuation of treatment due to either grade 3 or 4 treatment-related Adverse Event (AE) or a grade 2 treatment-related AE persisting for ≥ one month or recurring more than three times despite dose reduction.
* Patients must have adequate laboratory values:

  * Serum albumin ≥ 3g/dL
  * Aspartate Aminotransferase (AST)/Serum Glutamate Oxalacetate Transaminase (SGOT) and Alanine Aminotransferase (ALT)/Serum Glutamate Pyruvate Transaminase (SGPT) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to leukemic involvement
  * Serum bilirubin ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
  * Serum potassium, phosphorus, magnesium, and serum total calcium (corrected for serum albumin) or serum ionized calcium ≥ Lower Limit of Normal (LLN). Supplementation was allowed to correct potassium, calcium, and magnesium values prior to enrollment.
  * Thyroid Stimulating Hormone (TSH) and free Thyroxine (T4) within normal limits (WNL) (patients may have been on thyroid hormone replacement)
* Baseline measurement of left ventricular ejection fraction [assessment of the hearts ability to pump effectively]
* Assessment of patients ability to perform every day activities. Assessment by the Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.

Exclusion criteria:

* A candidate for hematopoietic stem cell transplantation
* Prior therapy with certain medications:

  * Therapeutic doses of sodium warfarin or any other anti-vitamin K drug (low doses for line patency were allowed).
  * Candidate for hematopoietic stem cell transplantation (HSCT)
  * Prior histone deacetylase (HDAC) inhibitor treatment of Chronic Myelogenous Leukemia (CML)
  * Concomitant use of drugs with a risk of causing QT complex (QTc) prolongation or torsades de pointes, CYP3A4/5 inhibitors, anti-cancer therapy or radiation therapy, valproic acid (within 5 days prior to study drug treatment or during the study), chemotherapy (within 3 weeks), immunotherapy (within 1 week), BCR-ABL kinase inhibitor ≤ 1 week of first treatment with panobinostat
* Patients who are in chronic phase chronic myeloid leukemia
* Impaired cardiac function or clinically significant cardiac diseases
* Concomitant use of drugs with a risk of possible risk of causing QTc prolongation or torsades de pointes
* Concomitant use of certain medications
* Impairment of Gastrointestinal (GI) function or GI disease
* Patients with unresolved diarrhea
* Women who are pregnant or breast feeding or women of childbearing potential not using an effective method of birth control
* Male patients whose sexual partners are women of child bearing potential not using effective birth control Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-02-23 (Actual); Primary Completion 2008-01-29 (Actual); Study Completion 2008-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (19):
  - City of Hope National Medical Center, Duarte, California
  - University of Colorado Health Sciences Center/Anschutz Cancer Pavilion, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Northwestern University Clinical Research Office, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University Chicago Hospital, Chicago, Illinois
  - Indiana Blood and Marrow Institute/St. Francis Hospital, Beech Grove, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hackensack University Medical Center/Oncology Research Dept., Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Emory University School of Medicine-Winship Cancer Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Clinical Trials Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Germany (7):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Munich

REFERENCES:
- [Result] Savelieva M, Woo MM, Schran H, Mu S, Nedelman J, Capdeville R. Population pharmacokinetics of intravenous and oral panobinostat in patients with hematologic and solid tumors. Eur J Clin Pharmacol. 2015 Jun;71(6):663-672. doi: 10.1007/s00228-015-1846-7. Epub 2015 May 5. PMID 25939707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 centers in 7 countries.
Pre-assignment Details: A total 27 Participants were enrolled in the study of which 27 participants discontinued the study treatment and 18 participants discontinued the study.
Period: Overall Study
Arm/Group | Panobinostat
Started | 27
Completed | 9
Not Completed | 18
Not completed — Disease progression | 12
Not completed — Death | 5
Not completed — New cancer therapy | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed in Full analysis set (FAS) population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study.
Groups:
- Panobinostat: Participants received panobinostat 20 mg orally OD, three times a week as part of a 4 week (28 day) treatment cycle. Panobinostat was administered at the same time each morning, and with an 8oz/240 ml of water after a fasting period of at least two hours (water was allowed). Participants could continue this treatment until an unacceptable toxicity that precludes further treatment was experienced, or until disease progression.
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22
  Black | 4
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Hematologic Response
Description: The primary efficacy variable was hematologic response, a composite endpoint defined as the overall of complete hematologic response (CHR), and of no evidence of leukemia (NEL) and of the return to chronic phase (RTC).
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed in Full analysis set (FAS) population was defined according to the intention-to-treat principle. Population included all participants enrolled into the study. Enrolled participant were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated because of a lack of evidence of activity in the targeted participant population.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Participants | 0

2. Secondary Outcome: Duration of Hematologic Response
Description: Duration of hematologic response is defined as the time from the first documentation of the hematologic response to the date of the first documentation of the disease progression
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. Enrolled patients were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated because of a lack of evidence of activity in the targeted Participant population. Because of a lack of evidence of hematologic response (primary objective), secondary efficacy endpoints were not analyzed.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Cytogenetic Response (CCyR) Rate
Description: Durations of complete cytogenetic response is defined as the time from the first documentation of the major/complete response to the first documentation of the disease progression.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

4. Secondary Outcome: Major (Complete/Partial) Cytogenetic Response Rate
Description: Durations of major/complete cytogenetic response is defined as the time from the first documentation of the major/complete response to the first documentation of the disease progression.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

5. Secondary Outcome: Complete Cytogenetic Response (CCyR) and Overall (Complete/Partial/Minor/Minimal) Cytogenetic Response (OCyR) Rates
Description: Cytogenetic response was assessed by bone marrow assessment based on the percentage of Ph+ metaphases by karyotype analysis on a bone marrow aspirate, was ideally assessed from a minimum of 20 metaphases in each bone marrow sample.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Major Cytogenetic Response
Description: The duration of response was defined as the time between the first documented response to the date of discontinuation due to progressive disease (PD) or death.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 2
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

7. Secondary Outcome: Major (MMR) and Complete (CMR) Molecular Response Rates
Description: Molecular response was defined as major (≤ 0.1% on the International Scale) and complete [absence of fusion gene of the BCR and ABL genes (BCR-ABL) on an quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay with a sensitivity of at least 4.5 logs below baseline].
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study. Enrolled patients were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated because of a lack of evidence of activity in the targeted Participant population. Due to insufficient data, this outcome could not be measured.
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

8. Secondary Outcome: BCR-ABL Mutations of Participants at Study Entry and, in Responding Participants and at the Time of Disease Progression
Description: A fusion gene of the BCR and ABL genes (BCR-ABL) messenger ribose nucleic acid (mRNA) expression (molecular response) was performed by quantitative polymerase chain reaction (qPCR) and mutational analysis was performed by direct sequencing technology, and both analyses were performed by Genzyme.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study. Enrolled participants were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated because of a lack of evidence of activity in the targeted Participant population.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Participants | 0

9. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressions free survival is defined as time between Day 1 cycle 1 and time to first documented disease progression or death. Disease progression will be determined as per response criteria.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 7
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Survival Time
Description: Overall survival time is defined as the time from the treatment start to the date of death due to any reason.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: as for outcome 7
Arm/Group | Panobinostat
Number analyzed (Participants) | 0

11. Secondary Outcome: Time to Peak Concentration (Tmax) of Panobinostat
Description: Tmax is defined as the time at which the Cmax occurs. It will be obtained from the Tmax parameter calculated by WinNonlin®. If there is no measurable Cmax in the subject's Pharmacokinetic (PK) profile, then Tmax will be missing for that subject. Tmax will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in Pharmacokinetic analysis set (PAS) population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Median (Full Range); unit: Hours
Groups:
- Panobinostat: Participants received panobinostat 20 mg orally OD, three times a week as part of a 4 week (28 day). Panobinostat was administered at the same time each morning, and with an 240 ml of water after a fasting period of at least two hours (water was allowed). Participants could continue this treatment until an unacceptable toxicity that precludes further treatment was experienced, or until disease progression.
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Hours
  Day 1: number analyzed (Participants) | 16
  Day 1 | 1.5 [0.2 to 3.4]
  Day 8: number analyzed (Participants) | 15
  Day 8 | 1.5 [1.0 to 3.4]

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Panobinostat
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations. It will be obtained from the Cmax parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Cmax will be missing for that subject. Cmax will be reported in units of ng/mL.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in PAS population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ng/mL
  Day 1: number analyzed (Participants) | 16
  Day 1 | 13.5 (7.0)
  Day 8: number analyzed (Participants) | 15
  Day 8 | 20.9 (15.0)

13. Secondary Outcome: Area Under the Plasma Concentration (AUC0-24) of Panobinostat
Description: Area under the curve (AUC) is defined as the area under concentration-time curve as a measure of drug exposure. The area under the plasma concentration-time curve from time zero to 24 hours.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 12
ng.hr/mL
  Day 1 | 139 (61)
  Day 8 | 148 (69)

14. Secondary Outcome: Last Observed Plasma Concentration (Clast) of Panobinostat
Description: Clast is defined as the Last observed (quantifiable) plasma concentration (Clast), in units of ng/mL. Blood samples were collected to assess Clast.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ng/mL
  Day 1: number analyzed (Participants) | 17
  Day 1 | 1.9 (2.4)
  Day 8: number analyzed (Participants) | 16
  Day 8 | 4.7 (8.2)

15. Secondary Outcome: Time of Clast (Tlast) of Panobinostat
Description: Time of Clast (Tlast) will be obtained from the Tlast parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Tlast will be missing for that participants. Tlast will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 12
Measure: Median (Full Range); unit: Hours
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Hours
  Day 1: number analyzed (Participants) | 17
  Day 1 | 23.9 [3.1 to 49.2]
  Day 8: number analyzed (Participants) | 16
  Day 8 | 24.1 [2.2 to 27.0]

16. Secondary Outcome: QT Interval (QTc) in Participants Receiving Oral Panobinostat at Baseline and Change From Baseline to Extreme Value
Description: QTc monitoring was performed on specified days (Cycle1: Day1, 5 and 26), as well as a single pre-dose ECG once weekly during Cycle1: Week2 and Week3, Cycle2, and all subsequent cycles. Patient eligibility was ensured by a screening QTcF interval calculated by eResearchTechnology(eRT) prior to the baseline assessments. Treatment decisions were based on QTc determined by the automated reading at the investigational site (commonly used the Bazett's correction,QTcB) or measured and calculated by trained personnel at the site. Dosing relied on the investigator's assessment of the 6 baseline ECGs (the average of the 6pre-dose QTc intervals) performed prior to Cycle1/Day1 dosing, of the 3pre-dose ECGs during Cycle1:Day5 and 26, and of the single pre-dose ECGs performed once weekly for the remaining weeks of Cycle1 and subsequent cycles. The Baseline and Change From Baseline to Extreme Value QTcF interval for analysis was calculated by eRT based on the 6 baseline ECGs obtained on Cycle1/Day1.
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study. Enrolled patients were those who had received at least one dose of study drug. The outcome measure was not achieved as the study was terminated because of a lack of evidence of activity in the targeted Participant population.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
ms
  Baseline: number analyzed (Participants) | 26
  Baseline | 396.6 (20.10)
  Change from Baseline: number analyzed (Participants) | 26
  Change from Baseline | 24.5 (9.58)

17. Secondary Outcome: Safety and Tolerability of Panobinostat
Description: Adverse Events (AE) are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Population: The analysis was performed on Safety population consisted of all participants who had received at least one dose of study medication and had one valid post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat
Number analyzed (Participants) | 27
Participants
  Participants with Adverse Events | 27
  Deaths | 16
  Serious Adverse Events | 13

ADVERSE EVENTS:
Time Frame: From Start of the Study up to Study Termination (approximately up to 18 Months).
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Arm/Group | Panobinostat
All-Cause Mortality (participants affected / at risk) | 16/27
Serious Adverse Events (participants affected / at risk) | 13/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Asthenia (General disorders) | 1
Catheter site haemorrhage (General disorders) | 2
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 4
Pneumonia (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=27)
Anaemia (Blood and lymphatic system disorders) | 10
Leukocytosis (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Tachycardia (Cardiac disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 7
Bacteraemia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
White blood cell count increased (Investigations) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes